CLINICAL TRIAL: NCT04700059
Title: Adaptation and Assessment of a Family Intervention Designed to Improve Maternal and Child Mental Health in a Resource-limited Setting
Brief Title: Family Intervention to Improve Maternal and Child Mental Health
Acronym: MCMH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Instituto Nacional Materno Perinatal (Unknown); Hospital San Bartolome (Other); AC PROESA (Unknown)
Responsible Party: Principal Investigator, Elizabeth Levey, MD, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB18-0533
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Adolescent Pregnancy
Keywords: Perinatal intervention; Intergenerational trauma
MeSH Terms: conditions — Historical Trauma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 10 perinatal home visits
  Interventions: Behavioral: Virtual perinatal home visiting
- Usual care (No Intervention): Routine medical care for mother and infant. Access to online resources.

INTERVENTIONS:
Behavioral: Virtual perinatal home visiting — 10 perinatal home visits
  Arms: Intervention

SUMMARY:
This pilot study will assess the acceptability, feasibility and efficacy of a family-based intervention to improve maternal and child mental health by increasing maternal sensitivity and decreasing offspring abuse among adolescent mothers in Perú, a middle-income country with high rates of childhood physical and sexual abuse, IPV, and adolescent pregnancy.

DETAILED DESCRIPTION:
Participants will be recruited from the prenatal clinics at INMP and San Bartolomé. Due to COVID-19, the prenatal clinics are currently conducting only telehealth visits. The interviews will be conducted using structured questionnaires that cover questions about socio-demographic characteristics, lifestyle characteristics, symptoms of depression or PTSD, history of trauma, and medical, obstetric and psychiatric history. Participants will be able to enter their responses online, with a research team member available to answer questions by phone, or they can give their answers by phone while a team member enters them. See attached Initial Questionnaire for details.

After the interview, each participant will be asked to provide the name of someone whom she anticipates will be helping her to care for the child. We expect that in most cases this will be a female relative of the participant, typically her mother or grandmother, but it may also be a friend or the baby's father. The participant will be given information about the study to provide to the other caregiver, and the interviewer will contact the other caregiver within a week of enrolling the participant and arrange for a convenient time for the caregiver to learn about the study and go through the informed consent procedures. If more than one person is providing significant support to the mother, she may identify up to two other caregivers. She can also identify a second caregiver at a later point.

Each participating family will be randomized to either the intervention arm or the usual care arm. Usual care consists of routine prenatal care and pediatric follow up at 2 weeks, 2 months, 4 months and 6 months. If enrolled prior to 20 weeks gestation, participants in both groups will receive a short phone call to check in every 4 weeks, until they reach 24 weeks gestation, to minimize the gap before the first visit at 28 weeks.

After delivery, obstetric records will be reviewed for information about gestational age, birth weight, and any complications. See attached Birth Data form for planned data collection.

Due to COVID-19, the intervention will begin with virtual visits conducting via videoconferencing. If, during the study period, it becomes safe to do home visits, we may switch to in-person home visits, or we may conduct the entire study with virtual visits. The intervention consists of 2 prenatal and 8 postpartum visits, with visit frequency gradually decreasing as mothers gain experience and confidence. Visits will last for up to 90 minutes to allow time for multiple caregivers to participate. Other caregivers will be encouraged to participate for the first 10 minutes and the last 20 minutes of the intervention sessions. As much as possible, visits will accommodate the family schedule, occurring at a time when all or most of the caregivers are at home. The perspectives of all caregivers will be elicited by the home visitor in order to facilitate a conversation among them about their preferences, concerns, and goals.

After completion of either the intervention or the control condition, the adolescent mothers will repeat the questionnaires about demographics, as well as anxiety, depression, PTSD and trauma history. If COVID-19 precautions are still necessary during this phase of the study, the post-intervention questionnaires will be completed in the same manner as the initial questionnaires, with data entered online with the support of the research team by phone. See attached Post-intervention Questionnaire for details. Interactions between the mother and infant, other caregiver and infant, and all three together will be video recorded and coded to assess caregiver sensitivity. If COVID-19 precautions are still necessary, these assessments will be conducted using video conferencing, and the video calls will be recorded and coded in the manner described. These recordings will be assessed and coded across five dimensions: "physical involvement," "verbal involvement," "responsiveness," "positive statements," and "control over child's activities," each rated 0-5 for the "quality" and "appropriateness" of caregiver behavior (Cooper et al., 2009; Farran, Kasari, Comfort, & Jay, 1986). Finally, the Still Face Paradigm will be conducted in which the mother-infant dyads will perform a video recorded 3-minute face-to-face interaction consisting of 1 minute normal, 1 minute still-face, and 1 minute reunion after still-face. Maternal behavior will be scored for sensitivity during normal and reunion phases (scored 0-5) (Murray, Fiori-Cowley, Hooper, & Cooper, 1996); infants will be scored for regulatory behavior (Braungart-Rieker, Garwood, Powers, & Wang, 2001; Murray & Trevarthen, 1985; Tronick & Weinberg, 1994) and dysregulated behavior, including gaze aversion, facial expression, crying, and agitated movement during each 1-second interval (Gunning, Halligan, & Murray, 2013).

We will record only what is necessary for the research record and take all steps necessary to blur/obscure the images of those who have not consented to the research and/or to being recorded or photographed. All interview guides and other study materials not currently available will be submitted to the IRB for approval prior to use.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be able to read and write Spanish.
* RCT will be limited to pregnant adolescents who are between the ages of 14-19 years and 12-34 weeks gestational age. Other caregivers (age 14 years or older) will be eligible if they are planning to be involved in infant care.
* Only pregnant adolescents receiving outpatient prenatal care at INMP or San Bartolomé will be approached as potential participants.
* Only pregnant adolescents who have been cleared by their attending doctor/nurse to engage in the approach/recruitment and interview procedure will be approached as potential participants.
* All infants born to adolescents enrolled during pregnancy will be eligible to be enrolled after birth.

Exclusion Criteria:

* Anyone unable to read and write Spanish.
* Any pregnant adolescent known to have a severe fetal anomaly will not be approached.
* Infants who are advised not to participate by their attending doctor or pediatrician.
* Children or adolescents who are wards of the state will not be enrolled.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Emotional availability scales | 6 months after birth
  Video recorded coded assessment of caregiver and infant interaction

SECONDARY OUTCOMES:
PHQ-9 | At enrollment and 6 months after birth
  Maternal depression
GAD-7 | At enrollment and 6 months after birth
  Maternal anxiety
PCL-C | At enrollment and 6 months after birth
  Maternal PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional Materno Perinatal, Lima, Peru

IPD SHARING:
Plan to Share IPD: No